CLINICAL TRIAL: NCT04548323
Title: Hypoalgesic Effects of Walking and Running Imagined in Sedentary Subjects and With High Levels of Physical Activity: A Prospective Cohort Study
Brief Title: Hypoalgesic Effects of Walking and Running Imagined
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Other Study IDs: uammadrid32
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Analgesia
Keywords: Motor imagery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Motor Imagery in Sedentary subjects
  Interventions: Behavioral: Motor imagery
- Motor Imagery active subjects
  Interventions: Behavioral: Motor imagery

INTERVENTIONS:
Behavioral: Motor imagery — Subjects will perform motor imagery tasks on the motor gestures of running and walking.

SUMMARY:
The main objective is to identify the hypoalgesic effect of the imagination of actions in sedentary subjects with high levels of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic participants
* men and women aged 18 to 65 years

Exclusion Criteria:

* insomnia
* nausea
* headache
* pregnancy
* use of painkillers in the last 24 hours
* presence of metal inside the head
* pacemaker
* wound on the area of electrodes' application
* drug consumption; (j) recent application of tDCS
* psychiatric disease impeding understanding of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects divided by their physical activity levels.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain pressure threshold | Change from baseline and immediately post-intervention
  Pressure Pain Threshold (PPT) is one of these tests and it is defined as the minimum force applied which induces pain. The measurement shall be carried out by using an algometer (pressure device that induces mechanical stimuli) is to standardize the amount of pressure applied in the neck region. The reliability of pressure pain thresholds according to raters or measurement frequencies is relatively high
Temporal sumation | Change from baseline and immediately post-intervention
  Temporal summation is a somatosensory measure that is performed by making small punctures in the area of interest.
Electrodermal activity | Change from baseline and immediately post-intervention
  Electrodermal Activity will be measured through the use of two electrodes that recorded changes in conductance through the skin located at the back of the dominant hand
Respiration Rate | Change from baseline and immediately post-intervention
  Respiration Rate will be measured through a pressure transducer located in the centre of the chest, where it was fixed by a strap.
Heart rate | Change from baseline and immediately post-intervention.
  Heart Rate will be measured by three electrodes located in the left area of the chest. One of the electrodes was placed in the middle zone while a second electrode was positioned on the lateral side, and a third one on the lower left side, below the first electrode.
Salivary stress | Change from baseline and immediately post-intervention.
  The Salivary Stress Test is a study that assesses fatigue and the type of stress (acute, moderate or chronic) presented by the subject.

SECONDARY OUTCOMES:
Visual and Kinesthetic Motor Imagery Ability | Change from baseline and immediately post-intervention
  Visual and Kinesthetic Motor Imagery Ability will be measured with Movement Imagery Questionnaire-Revised (MIQ-R). MIQ-R has four movements repeated in two subscales, a visual and a kinesthetic one. Additionally, a score between 1 and 7 is assigned, with 1 representing difficulty in picturing the motor image or difficulty in feeling the movement previously made, and 7 representing the maximum ease. The internal consistencies of the MIQ-R have been consistently adequate with Cronbach's α coefficients ranging above 0.84 for the total scale, 0.80 for de visual subscale and 0.84 for the kinesthetic subscale.
The degree of physical activity | Immediately before the intervention.
  The degree of physical activity was objectified through the The International Physical Activity Questionnaire (IPAQ) questionnaire, which allows the subjects to be divided into three groups according to their level of activity, which can be high, moderate, and low or inactive. The IPAQ consists of 7 questions about the frequency, duration and intensity of activity (moderate and intense) performed in the last seven days, as well as walking and sitting time on a workday. The IPAQ scoring protocol assigns the following MET values to walking, moderate, and vigorous intensity activity: 3.3 METs, 4.0 METs, and 8.0 METs, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain